CLINICAL TRIAL: NCT04518098
Title: Feasibility and Efficacy of the Remotely Delivered STABLE Program for Community-dwelling Older Adults With Cancer: A Randomized Controlled Feasibility Trial
Brief Title: STABLE (Strength Training and Balance Leg Exercise) Study
Acronym: STABLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Schroder Sattar, Assistant Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BIO-1396
Record Dates: First submitted 2019-07-18; First posted 2020-08-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Neoplasms
Keywords: resistance and balance training; fall prevention; older adults; cancer; Exercise
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors who collect outcome data will be blinded to group allocation. Participants will be advised to refrain from disclosing their group allocation to the outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the IG will receive the STABLE intervention, which entails orientation, and undertaking a remotely delivered resistance and balance training regimen 3 times weekly for 3 months
  Interventions: Other: Strength and balance exercise
- Control group (No Intervention): Participants in the CG will not receive the intervention, and will be advised to carry out their usual daily activities.

INTERVENTIONS:
Other: Strength and balance exercise — The exercise program consists of muscle strengthening and balance training exercises that progress in difficulty. After completion of the baseline assessment and randomization, IG participants will receive orientation and learn the exercise routines (in the Cancer Rehabilitation Clinic within the Faculty of Rehabilitation Medicine at the University of Alberta). The duration of training is 3 months (40-50 minutes per scheduled session, three times a week) at home, with a minimum of one live group session supervised by the CEP, a minimum of one independent home session supported by the Active Living module of the HEAL-ME application; (the third session can be a live session or independent session at the participant's discretion).
  Arms: Intervention group

SUMMARY:
Falls are a major health concern amongst older adults with cancer, and are often related to decreased physical strength due to effects of cancer and its treatments. Ample evidence demonstrates the benefits of exercise programs incorporating strength and balance training on lower body strength, balance, and fall prevention older adults. However, gaps in research exist within the geriatric oncology context. The purpose of this study is to determine the feasibility and efficacy of a 3-month, remotely delivered exercise program regimen on lower body strength, balance, and falls in older adults with cancer.

This observer-blinded, randomized controlled feasibility trial aims to recruit older cancer patients (aged ≥65). Participants in the intervention group will undertake the exercise program 3 times weekly for three months. Data collection will include sociodemographic survey, baseline, end-of-intervention (3-month) assessment, follow-up (6-month) assessment, chart review, and exit survey. Descriptive and inferential statistics will be used to analyze data, following the intention-to-treatment principle.

Data generated from this research project will inform design of a subsequent, larger exercise intervention trial. This is an important step to establish the knowledge base regarding provision of exercise interventions as a fall prevention strategy to reduce falls and their negative outcomes in older patients in the community.

DETAILED DESCRIPTION:
Hypothesis: A remotely delivered, 3-month resistance and balance training program will result in an increase in lower body strength, improvement in balance, as well as a lower fall rate compared to control. This is important because of the potential to improve quality of life for older adults with cancer, decreasing societal and economic costs associated with injuries and injury-related treatment and hospitalizations, and avoiding unnecessary modifications to cancer treatment.

Objectives

1. Determine the feasibility of a remotely delivered resistance and balance training program over a 3-month period in community-dwelling older adults (≥65 years of age) who have undergone or are receiving systemic cancer treatment; and
2. Explore the efficacy of this exercise program on lower body strength, balance, and fall rates and obtain estimates to inform the design of a larger randomized controlled trial.

METHOD:

The STABLE (Strength Training And Balance Leg Exercise) study is an observer-blinded, parallel group (IG vs. CG) randomized controlled trial. Participants Study participants will be recruited over a 12-month period from the cohort of older patients with cancer referred to the Cross Centre Institute, Edmonton, Alberta.

Sample size determination:

Assuming three covariates (age, gender, and cancer stage), a correlation of 0.95 between repeated measures, based on an effect size of 0.68 in our pilot study, and a significance level of 5%, we estimate a sample size of 37 participants in each group would have 80% power to detect differences between and within the control and treatment groups. Using Bonferroni's Correction for Multiple Comparisons, to allow for an adherence rate of 90% throughout the study and an overall attrition rate of 3%, 74 participants in total are required in both the control and treatment groups.

Procedure:

Information about the study (with contact information) will be provided to clinicians at the Cross Cancer Institute to disseminate to patients. Posters will also be placed in waiting areas of oncology clinics and chemo infusion clinics. Patients who are interested may choose to contact study staff to learn more about the study. At the time of informed consent, all participants will be asked whether they have a computer or a tablet-styled device (e.g. iPad), those who do not will be provided with an iPad (on loan during the intervention), for the duration of the study. The informed consent process will also include obtaining participants' permission to collect information from their medical chart, including comorbidities, cancer type, stage, and treatment intent and type.

Randomization:

After informed consent and collection of baseline data, randomization will take place. The randomization will be performed through the Research Electronic Data Capture [RedCap7.1.1] database system. Participants will be stratified by treatment status (on/off systemic therapy) and then randomized into parallel groups with a 1:1 allocation ratio to either IG or CG.

Blinding:

Single blinding will be applied by the independent assessor who conducts the outcome assessment as well as the statistician who will carry out the statistical analyses. Instructions and reminders will be provided to participants to avoid disclosing their group allocation to the outcome assessor prior to each assessment appointment.

Adverse events Exercise trials in older adults with cancer have been found to be safe, and adverse events are rare. Therefore, we anticipate a low adverse event rate for this study. Any adverse events during the training sessions will be documented and graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4. In the rare event of an adverse event, the participant's treating physician will be notified.

Equipment:

The equipment required for the strength and balance training will include exercise bands of various resistance levels, all of which will be provided to the IG participants for use free of charge. iPad devices will be provided to participants on loan to use during the study period.

Intervention:

Intervention is described in section below.

Progression:

Each IG participant's exercise performance will be monitored closely by the CEP, and exercise loads and/or progressions will be titrated accordingly during each exercise session. Progression of balance training will occur by graduating from holding onto a stable structure to performing the exercise independent of support. For the resistance-training component, once the participant can complete all of the highest number of prescribed repetitions for all of the sets of an exercises with a given resistance band, she/he will progress to the next level of resistance band for the subsequent workout. The increase in resistance will result in dropping the repetitions performed to the lower range of the prescribed repetition zone with the goal of increasing number of repetitions performed until the upper limit of the prescribed repetition zone is once again achieved.

Control:

The Control Group (CG) will not receive the intervention, and will be advised to carry out their usual daily activities. As mentioned, data collection for CG participants will occur at baseline and at 3- and 6-month follow-up by an independent assessor blinded to study group allocation.

Data management:

All collected data will be managed through a password-protected, secure database (RedCap7.1.1) Files containing participant information will be de-identified and stored in a locked cabinet at the site PI's office at the University of Alberta.

Assessments:

Outcomes will be measured at baseline: t0, prior to starting the STABLE program), 3 months (t1, when the intervention period is complete), and at 6 months (t2, to provide a longitudinal perspective of the outcome measures; specifically, stabilization of gains). After informed consent, participants will complete the baseline assessment, which will include a survey (sociodemographic information, functional status, fall history, fall efficacy).

Baseline assessment will also assess lower body strength/balance, and history of falls. During the 3-month follow-up period, falls in IG participants will be assessed weekly via built-in questions on the App, and falls in CG participants will be assessed weekly either online or by weekly phone calls based on participant preference.

The 3-month assessment entails assessment of both groups for lower body strength, balance, falls, as well as update on clinical data, fall-efficacy, and functional status to provide context. For IG participants, 3-month data collection will also include an exit survey to collect participants' opinions regarding the intervention, any difficulties related to exercising and adherence, as well as feedback for future improvement. This survey will be scheduled separately and administered by the research assistant to ensure continual blinding of the outcome assessor.

The 6-month follow-up assessment will collect data from both groups on lower body strength, balance, and falls, as well as functional status and fall efficacy.

All outcome assessments will be carried out by an independent assessor blinded to group allocation and not involved in analysis of study results.

Adherence, retention, and concomitant care:

Time will be allocated during each group session to promote adherence and provide opportunity to ask questions. Additionally, during each exercise session, participants will also be encouraged by the CEP to carry out the full set of routines as prescribed. Participants who report falls will be asked about circumstances of their falls (as per the recommendations of the AGS/BGS), and will be referred for appropriate follow-up.

Outcome Measures are described in section below.

STATISTICAL ANALYSIS:

Standard principles for RCTs will be followed for statistical analysis (e.g. including performing of sensitivity analysis for non-ignorable missing data). Descriptive statistics (e.g. means, standard deviations, counts, percentages) will be used to describe patient characteristics (i.e. age, sex, gender, number of comorbidities and medications, cancer site, stage, treatment type) as well as use of mobility aid, functional status, and fall efficacy. Descriptive analysis will be used to summarize each group for primary and secondary outcomes (frequencies, means, SDs, medians, IQRs, 95% CIs). Data will be assessed for normality before inferential statistics will be conducted. To avoid bias in estimating the intervention effect, an intention-to-treat analysis will be performed (i.e., inclusion of all measures in all participants irrespective of whether they completed the intervention).

To answer Research Question 1: What is the feasibility of this 3-month exercise program, in terms of recruitment, retention, adherence, outcome capture, completion, and acceptability? Descriptive statistics (numbers and proportions) will be used to analyze recruitment rate, retention, adherence, outcome capture, and completion (based on entire sample and gender). Data from exit surveys will be summarized to determine satisfaction with study procedures and participation experience and what could be improved for participants in larger trial.

To answer Research Question 2: What are the preliminary effects of a 3-month strength and balance exercise on lower body strength, balance, and fall rates in community-dwelling older adults with cancer? We will build generalized linear mixed-effect models to perform a longitudinal analysis of our lower body strength, balance, and falls outcomes, respectively. Advantages of using generalized linear mixed-effect models are they can model repeated measures using a variety of correlation structures and also provide parameter estimates when data are missing. We will build our models for each of the three outcomes-lower body strength, balance, and falls, as follows. To characterize time-dependent changes in an outcome, we will include time as both a fixed effect and a random effect (second-level effect). We then will add the study group variable into the model to determine the unadjusted associations between the study group variable and the outcome variable. To adjust these associations for the effects of our covariates (i.e., age, sex, cancer stage), we then will add all of the covariates into the models. In this adjusted model, a parameter estimate will be considered significant if p<0.05. We will also reference the minimum clinically important difference (MCID) or substantial meaning change values for the primary outcomes (i.e., 2 repetitions for the 30 seconds chair stand and improvement of ≥1 point for the balance test). Additionally, we will also perform an exploratory analysis on other variables (i.e. functional status, treatment exposure) to determine possible associations with three study outcomes.

Ethics approval:

Ethics approval has been granted by the Research Ethics Boards of the University Saskatchewan and is being sought from the Health Research Ethics Board of Alberta: Cancer Committee. Operational approval will be sought from the Cross Centre Institute and Alberta Health Services. During the informed consent process, participants will be informed that they can withdraw from the study at any time and, if they choose to stop participating, data collected up to the point of their withdrawal will be included in the data analysis; however, no further data will be collected.

ELIGIBILITY:
Inclusion criteria:

* Adults aged 65 or above;
* living in the community;
* have a confirmed diagnosis of any stage of lung, breast, prostate, or colorectal cancer; - currently receiving, starting or have completed systemic anti-cancer therapy;
* life-expectancy of at least 9 months (in consideration of the measurement period of the study and also avoid burdening patients who are near the end-stage of their disease); and - completed the PAR-Q screening or have approval of their treating physician.

Exclusion criteria:

* presence of brain metastases;
* presence of unstable metastases as per treating physician (e.g., bone metastasis in a weight-bearing area, recent bone fracture);
* presence of any conditions that would potentially interfere with their ability to carry out the exercise interventions (e.g., mobility impairment, poorly controlled pain, severe vision/hearing loss, severe arthritis that limits ambulation, left-sided heart failure, neurological or musculoskeletal conditions);
* self-reported history of light-headedness during physical activities; syncopal episodes within the past month; and
* participation in any form of structured exercise program (that are at least 30 minutes per week) at the time of consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
30-second Chair Stand test | Baseline, 3 & 6 months - to measure change
  The 30-second chair stand test will begin with having the participating sitting upright in the middle of the chair with arms folded across the chest with hands placed on the front of the opposite shoulder. The feet are placed flat on the ground at shoulder width and slightly behind the knee. At the initiation of the test using a count down of "ready…go," the participant will stand upright (knees straight and torso fully erect) while maintaining the hand position on the shoulder and then return to a fully seated position in which body weight is shifted from the feet to the chair. The participant will complete as many stand-sit cycles as possible in the 30-second period. The number of sit-to-stands completed within the 30 seconds will be recorded and interpreted based on age group and gender as recommended by the Centers for Disease Control and Prevention STEADI guideline.
Balance test | Baseline, 3 & 6 months - to measure change
  Static balance ability will be measured using the Side-by-side Stand (SBS), Semi-tandem Stand (ST), and Full tandem Stand (FT). Participants will be asked to maintain their balance in the three different positions. The amount of time they succeed in maintaining the various positions, in seconds, will be recorded based on the following criteria: Side-by-side 10 sec, semi-tandem 10 sec (1 point); tandem 10 sec (2 points), tandem 3-9.99 second (1 point).
Fall assessment | Baseline, 3 & 6 months - to measure change
  Falls will be assessed at t0, t1, and t2 as described, by self-report following recommendations of fall assessment as outlined by the American Geriatrics Society/British Geriatrics Society (AGS/BGS)

CONTACTS AND LOCATIONS:
Overall Officials: Schroder Sattar, RN, PhD, Principal Investigator — College of Nursing; Margaret McNeely, PhD, Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sattar S, Haase KR, Alibhai SMH, Penz K, Szafron M, Harenberg S, Amir E, Kuster S, Pitters E, Campbell D, McNeely ML. Feasibility and efficacy of a remotely delivered fall prevention exercise program for community-dwelling older adults with cancer: Protocol for the STABLE trial. J Geriatr Oncol. 2022 Nov;13(8):1273-1280. doi: 10.1016/j.jgo.2022.06.009. Epub 2022 Jul 2. PMID 35792037